CLINICAL TRIAL: NCT01411202
Title: Outpatient Pleurodesis Using Sclerosants(OPUS):Comparing Doxycycline Pleurodesis to Continued Drainage With the Pleurx Catheter System in the Treatment of Malignant Pleural Effusions in the Outpatient Setting
Brief Title: Effectiveness of Doxycycline for Treating Pleural Effusions Related to Cancer in an Outpatient Population
Acronym: OPUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008362-01H
Record Dates: First submitted 2011-06-13; First posted 2011-08-08 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Malignant Pleural Effusion
Keywords: Malignant Pleural Effusion; Doxycycline; Pleurodesis; Pleurx catheter
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Doxycycline; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Experimental): Pleurx insertion with injection of 500mg of doxycycline in 50cc of normal saline.
  Interventions: Drug: Doxycycline
- Normal Saline (Placebo Comparator): Pleurx insertion with placebo injection of 50cc of normal saline
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Doxycycline — One time injection 500mg of powdered doxycycline reconstituted with 50cc of normal saline via Pleurx catheter
  Arms: Doxycycline
Other: normal saline — One time injection of normal saline (placebo) into Pleurx catheter
  Arms: Normal Saline

SUMMARY:
Patients with cancer may experience problems with their breathing due to a fluid accumulation around their lungs called malignant pleural effusion (MPE). This fluid can be drained but draining may not stop the fluid from accumulating again. MPE can cause shortness of breath during activity and at rest leaving patients feeling as though they cannot catch their breath enough to be comfortable. Other symptoms can include pain, cough and weight loss.

One way to stop the fluid from accumulating is to create scar tissue between the lung and chest wall so there is no more room for fluid accumulation. This procedure is called pleurodesis. Pleurodesis is the standard of care at most centres across Canada. This procedure is done by injecting a drug into the space between the lung and chest wall through a catheter, Doxycycline is one of the drugs currently used for this purpose. Traditionally, patients are admitted for pleurodesis, mostly because the size of the catheter used to inject the medication is very large but also because of the potential complications that can happen with these larger chest tubes.

At our centre, most patients with MPE are managed at home with a smaller sized catheter known as a Pleurx catheter. The Pleurx catheter allows patients to remain at home for treatment and trained staff come into the home to both drain the MPE and monitor the patient. Sometimes, patients experience pleurodesis through use of the Pleurx catheter alone.

Pleurodesis with doxycycline can happen faster than with the Pleurx catheter alone. It has been our experience with a limited number of patients that it is safe to perform pleurodesis using the Pleurx catheter for doxycycline injection in an outpatient setting.

DETAILED DESCRIPTION:
Malignant pleural effusions (MPE) occur in 25 - 50% of malignancies, represent advanced disease and carry with it significant morbidity. It is estimated that 75% of malignant effusions are symptomatic at the time of presentation, with dyspnea being the most common complaint. Cough, weight loss and chest pain may also be presenting symptoms. The diagnosis of MPE often carries with it a poor prognosis with an average survival of 3-9 months. Thus, management of MPE is generally palliative, aimed at alleviating the associated symptoms, while incurring minimal discomfort and disruption of patients activities of daily living. Limiting the number of days spent hospitalized ia also a consideration. Currently, the most common treatment for MPE involves tube thoracostomy and pleurodesis using a sclerosing agent. Use of Doxycycline as a sclerosing agent has been shown to be both safe and efficacious with only minor complications. Traditionally, pleurodesis with Doxycycline has been performed in the inpatient setting.

The Pleurx catheter (Cardinal Biomedical) is the only small bore catheter commercially available that has been specifically designed for long term indwelling drainage of MPE. In order to reduce the chance of dislodgement and minimize infection rates, it is tunnelled under the skin for approximately 5 cm before entering the pleural space. These indwelling catheters can provide excellent symptom control and have also been associated with spontaneous pleurodesis rates comparable to many chemical pleurodesis rates.

Pleurx has been compared to inpatient doxycycline pleurodesis via chest tube with no difference in survival, safety or efficacy noted. However, hospital stay was significantly shorter in the Pleurx group, 1 day versus 6.5 days.

The aim of this study is to determine the effectiveness of outpatient pleurodesis, using doxycycline administered via Pleurx catheter. This will be a randomized clinical trial comparing the time to pleurodesis in patients with malignant pleural effusion receiving doxycycline + Pleurx catheter versus Pleurx catheter alone.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of symptomatic and moderate sized (>1/3 of hemithorax) MPE
2. Persistent malignant pleural effusion that is free-flowing
3. Symptomatic improvement after therapeutic thoracentesis
4. Life expectancy of at least three months (duration of study follow-up)
5. 90% radiographic apposition of parietal and visceral pleura
6. Residence within 30 minute radius from The Ottawa Hospital

Exclusion Criteria:

1. Previous lobectomy or pneumonectomy on affected side
2. Multiple loculations
3. Trapped or entrapped lung
4. Untreated pleural infection
5. Abnormal coagulation profile (INR>1.5 and / or platelet count <50 x 10*9/L)
6. Planned intrapleural chemotherapy (however participants may receive concomitant systemic chemotherapy, mediastinal radiation therapy or steroids)
7. Life expectancy less than 3 months
8. Multiple co-morbidities limiting out-patient management of pleural effusion
9. Tetracycline / Doxycycline allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-06; Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to pleurodesis | up to 90 days post PleurX insertion
  measured in days after Pleurx catheter insertion up to 90 days

SECONDARY OUTCOMES:
Pleurodesis rates at 90 days post Pleurx insertion | 90 days post Pleurx insertion
  defined by the BTS guidelines, where complete pleurodesis is defined as lack of fluid re-accumulation, allowing for removal of the pleural catheter. Failed pleurodesis is defined as re-accumulation of fluid and symptoms requiring repeated pleural procedures
Number of participants with adverse events | 90 days post Pleurx insertion
  Most common complications include: pleural infection / cellulitis, pain, catheter obstruction and symptomatic loculated effusion. Other adverse events will also be collected.
Effects on pulmonary function | 90 days post Pleurx insertion
  Pulmonary Function testing will be performed prior to and post PleurX catheter insertion and prior to each follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: K. Amjadi, MD, FRCPC, Principal Investigator — Ottawa Hospital
Locations (2):
- Canada (2):
  - Ottawa Hospital, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Undecided